CLINICAL TRIAL: NCT01023490
Title: A Randomised, Double-blind, Placebo-controlled Study to Check Whether Vitamin D Will Lead to a Decrease in Pain Intensity in Patients Suffering From Chronic Pain and Hypovitaminosis D
Brief Title: Vitamin D Treatment to Patients Suffering From Chronic Pain and Vitamin D Hypovitaminosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TASMC-09-SB-0494-CTIL
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Back Pain; Hypovitaminosis D
Keywords: back pain; hypovitaminosis D
MeSH Terms: conditions — Back Pain; Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Vitamin D (Active Comparator): 34,500 IU vitamin D per week
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — 34,5000 IU vitamin D per week
  Arms: Vitamin D
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to check whether vitamin D will lead to a decrease in pain intensity compare to placebo, in patients suffering from chronic pain.

DETAILED DESCRIPTION:
Vitamin D is a complex nutrient that functions as a hormone to benefit numerous body tissues.

Vitamin D is naturally produced by skin exposed to ultraviolet B. Despite the fact that Israel is a sunny country, a majority of all patients, and particularly those with pain, have inadequate intake of vitamin D.

Vitamin D therapy is easy for patients to self administer, well tolerated, and very economical.

In this study, we'll check whether vitamin D will lead to a decrease in pain intensity in patients suffering from chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* men and women over 18, who suffer from chronic pain and hypovitaminosis D

Exclusion Criteria:

* patients that are treated with vitamin D

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The objective of this study is to check whether vitamin D will lead to a decrease in pain intensity compare to placebo, in patients suffering from chronic pain. | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Pain Medicine Unit, Tel Aviv, Israel